CLINICAL TRIAL: NCT02953106
Title: Proof of Concept Study to Assess Downstream Effects of Using Combined Intranasal Fluticasone Propionate Plus Azelastine Nasal Spray on Asthmatic Inflammation in Patients With Persistent Asthma and Allergic Rhinitis
Brief Title: Effects of Intranasal Fluticasone Plus Azelastine on Airway Inflammation in Patients With Asthma & Allergic Rhinitis
Acronym: MAN06
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The company providing study IMP was unable to supply further batches of IMP.
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-001093-17
Record Dates: First submitted 2016-10-28; First posted 2016-11-02 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Asthma, Allergic; Rhinitis,Allergic; Allergy
Keywords: Asthma; Rhinitis; Dymista; allergy
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Hypersensitivity; Rhinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azelastine-Fluticasone Nasal (Active Comparator): 137 micrograms azelastine hydrochloride / 50 micrograms fluticasone propionate per actuation. 1 squirt twice daily
  Interventions: Drug: Azelastine-Fluticasone Nasal
- Placebos (Placebo Comparator): contains the same components as Dymista nasal spray with the exception of the active ingredients. 1 squirt twice daily.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Azelastine-Fluticasone Nasal — 137 micrograms azelastine hydrochloride / 50 micrograms fluticasone propionate
  Other Names: Dymista
  Arms: Azelastine-Fluticasone Nasal
Drug: Placebos — Placebo nasal spray
  Arms: Placebos

SUMMARY:
Single centre, double-blind, placebo controlled, adaptive design, cross-over trial. The primary objective is to assess the additive effects of using combined intranasal fluticasone propionate plus azelastine nasal spray on airway hyperresponsiveness. This is in patients with persistent asthma and allergic rhinitis, receiving inhaled steroid.

DETAILED DESCRIPTION:
The unified allergic airway describes patients who have both asthma and allergic rhinitis. Both conditions have similar underlying pathophysiology in terms of T-helper 2 (Th2) cell activation. Patients with unified allergic airway disease have a greater burden in terms of impaired quality of life, and the presence of airway hyper-responsiveness (AHR) to methacholine is a hallmark of their underlying asthmatic inflammatory process. Targeting the Th2 allergic airway with a topical antihistamine may improve airway hyperresponsiveness.

It has previously been shown that in patients with unified allergic airway disease, using inhaled fluticasone alone (100 micrograms per day) produced a 1.2 doubling dilution (dd) shift in the provocative concentration of methacholine required to reduce forced expiratory volume (FEV1) by 20% (PC20). However when adding nasal fluticasone to the inhaled steroid, there was a 1.79 dd shift. This difference (0.58 dd, 95% CI 0.78, 1.95) was not statistically significant. However the combined treatment did result in significant improvement in rhinitis quality of life, nasal inflammation and inspiratory flow.

The investigators will repeat this previous concept, but compare intranasal fluticasone with azelastine (an antihistamine) nasal spray versus placebo nasal spray, in atopic asthmatic patients on inhaled steroid. This will be to assess effects on methacholine PC20, the primary outcome, and to assess the effects on the following secondary outcomes: Exhaled nitric oxide (FeNO), FEV1, morning peak expiratory flow (PEF), impulse oscillometry, peak nasal inspiratory flow (PNIF), nasal nitric oxide (NO), blood eosinophils, eosinophilic cationic protein (ECP), nasal symptoms, asthma control and quality of life; and rhinitis quality of life.

Twenty adults 18 and up, with allergic asthma will be enrolled. They will have a run-in on 2 weeks of 200 micrograms beclometasone inhaler and then be randomised to add either intranasal fluticasone and azelastine, or placebo nasal spray to their treatment (double blind). Treatment period one will be 3-5 weeks followed by a washout of 2-4 weeks, and crossover to treatment period two for 3-5 weeks. Due to the crossover nature of this study participants will receive both treatments in random order. There will be an Interim analysis after 20 participants complete the study per protocol and the exact required sample size will be recalculated (Pocock/adaptive design).

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, aged 18 years and above, with persistent asthma and allergic rhinitis
* On a minimum of 200μg BDP of Inhaled corticosteroid (ICS)
* FEV1 ≥ 60 % predicted
* Positive skin prick test, or record of elevated allergen-specific IgE to at least 1 perennial allergen
* Methacholine PC20 < 8mg/ml at Visit 1
* Ability to give informed consent

Exclusion Criteria:

* Other respiratory diseases such as COPD, bronchiectasis or allergic bronchopulmonary aspergillosis (ABPA) which are considered to be significant in the opinion of the study physician Nasal polyps ≥ Grade 2
* An asthma exacerbation or respiratory tract infection requiring systemic steroids and/or antibiotics within 1 month of the study commencement, or 3 months if hospital admission was required
* Any clinically significant medical condition that may endanger the health or safety of the participant. For example: Patients who have tuberculosis or any type of untreated infection or have had recent surgical operation or injury to the nose or mouth.
* Participation in another trial within 30 days before the commencement of the study
* Pregnancy or lactation
* Unable to comply with the procedures of the protocol
* Unable or unwilling to consent
* Taking prohibited medications as listed in section 6.7.2 Prohibited Medications
* Hypersensitivity to the active substances or to any of the excipients of Dymista Nasal Spray.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Methacholine PC20 | 3-5 weeks
  The provocative concentration of methacholine required to produce a 20% drop (PC20) in forced expiratory volume in 1 second (FEV1)

SECONDARY OUTCOMES:
Exhaled nitric oxide (FeNO) | 3-5 weeks
  A measurement of the amount of inflammation in the airways
Forced expiratory volume in 1 second (FEV1) | 3-5 weeks
  The amount of air exhaled in the first second of a forced expiration.
Morning peak expiratory flow (PEF) | 3-5 weeks
  A measurement of how quickly a patient can blow air out of their lungs
Airway resistance at 5Hz (R5) | 3-5 weeks
  A measurement of the total airway resistance at the frequency of 5 Hertz
Airway resistance at 20Hz (R20) | 3-5 weeks
  A measurement of the proximal airways resistance at the frequency of 20 Hertz
Peripheral airway resistance (R5-R20) | 3-5 weeks
  A measurement of the peripheral airway resistance by taking the resistance at 5Hz and subtracting the resistance at 20 Hertz
Airway Reactance (X5) | 3-5 weeks
  A measurement of the peripheral capacitive reactance at the frequency of 5 Hertz
Airway Reactance area under the curve (AX) | 3-5 weeks
  A measurement of the reactance area between the negative reactance trend and zero.
Domiciliary peak nasal inspiratory flow (PNIF) | 3-5 weeks
  A measurement of how open or blocked the nasal passages are.
Nasal nitric oxide (NO) | 3-5 weeks
  A measurement of the amount of inflammation in the nasal passages.
Blood eosinophils | 3-5 weeks
  A measurement of the amount of eosinophils in the blood
Eosinophilic cationic protein (ECP) | 3-5 weeks
  A measurement of the amount of Eosinophilic Cationic Protein (ECP) in the blood
Total nasal symptom score (TNS4) | 3-5 weeks
  A questionnaire to assess four (4) types of nasal symptoms: runny nose, blocked nose, itchy nose, and sneezing.
Asthma control questionnaire (ACQ) | 3-5 weeks
  A questionnaire to measure the degree of a person's asthma control
Asthma quality of life questionnaire (AQLQ) | 3-5 weeks
  A questionnaire to measure the functional problems that are most troublesome to adults with asthma.
Rhinitis quality of life questionnaire (RQLQ) | 3-5 weeks
  A questionnaire to measure the functional problems that are most troublesome to adults with rhinitis.
Visual analogue scale (VAS) | 3-5 weeks
  a 10 cm line horizontal describing rhinitis symptoms. zero being "not bothersome" and ten being "very bothersome".

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lipworth, MD, Principal Investigator — Scottish Centre for Respiratory Reseach
Locations (1):
- Scottish Centre for Respiratory Research, University of Dundee, Ninewells Hospital and Medical School, Dundee, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No